CLINICAL TRIAL: NCT02842203
Title: Use of ctDNA for Monitoring of Stage III Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Schoen, Professor of Medicine & Epidemiology, University of Pittsburgh
Other Study IDs: STUDY19070371; U01CA152753 (NIH)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Stage III Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples; formalin-fixed, paraffin-embedded tumor blocks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will evaluate circulating tumor DNA (ctDNA) as a prognostic marker and as a monitor of disease recurrence in stage III colorectal cancer (CRC).

DETAILED DESCRIPTION:
Circulating tumor DNA (ctDNA) are small fragments of nucleic acid that originate from apoptotic or necrotic tumor cell turnover. Characteristic of the malignant process, ctDNA can be assessed in plasma and offers the potential of a sensitive and specific biomarker for prognostic information on disease-free or overall survival, and predictive information on chemotherapy resistance and probability of lack of response to treatment. This study will evaluate ctDNA as a prognostic marker and as a monitor of disease recurrence in stage III colorectal cancer (CRC). We will recruit newly diagnosed stage III CRC patients, determine their tumor mutational profile, and systematically collect high volume (>10 ml), serial plasma specimens every 3 months for up to 3 years and every 6 months in years 4-5 for ctDNA and concurrent carcinoembryonic antigen (CEA) measurement. Clinical outcome and survival will be tracked. The resulting data will permit assessment of ctDNA as a prognostic marker for disease-free and overall survival and as a monitor of disease recurrence in comparison with CEA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with CRC Stage III A, B, or C
* Age ≥18 years
* Willingness to provide blood samples for research purposes
* Ability to understand written informed consent document, and written informed consent provided

Exclusion Criteria:

* Blood sampling would compromise patients overall health such as presence of severe anemia
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present in a UPMC Cancer Center and meet the criteria for this study will be approached by their treating physician about participation.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
ctDNA assessment and relation to clinical outcome | up to 5 years
  The relationship between ctDNA and survival (both progression-free and overall) will be evaluated. Both the total load of ctDNA and the specific mutation(s) identified will be evaluated.

SECONDARY OUTCOMES:
ctDNA versus CEA | up to 5 years
  ctDNA predictors of outcome will be compared to CEA

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schoen, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available according to NIH data sharing policies.
Time Frame: De-identified individual participant data will be made available according to NIH data sharing policies.
Access Criteria: De-identified individual participant data will be made available according to NIH data sharing policies.

REFERENCES:
- [Derived] Borhani AA, Zhang P, Diergaarde B, Darwiche S, Chuperlovska K, Wang SC, Schoen RE, Su GL. Role of tumor-specific and whole-body imaging biomarkers for prediction of recurrence in patients with stage III colorectal cancer. Abdom Radiol (NY). 2025 May;50(5):1907-1915. doi: 10.1007/s00261-024-04656-3. Epub 2024 Nov 2. PMID 39487920